CLINICAL TRIAL: NCT05067114
Title: Solutions for Atrial Fibrillation Edvocacy (SAFE) Improving Awareness and Access to Atrial Fibrillation Screening for Detection and Referral for Treatment
Brief Title: Solutions for Atrial Fibrillation Edvocacy (SAFE)
Acronym: SAFE
Status: Completed | Type: Observational
Sponsor: American Pharmacists Association Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 021
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cardiovascular Diseases; Cardiac Arrhythmia; Atrial Fibrillation
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: Screening, detection, and referral for atrial fibrillation
  Interventions: Device: Screening, detection and referral for atrial fibrillation

INTERVENTIONS:
Device: Screening, detection and referral for atrial fibrillation — In-pharmacy cardiovascular risk assessment plus AliveCor KardiaMobile reading

SUMMARY:
The aim of this demonstration project is to create an additional access point in the community at local pharmacies for atrial fibrillation screening, detection, and referral to physicians for follow-up and initiation of evidence-based therapy when appropriate.

DETAILED DESCRIPTION:
The APhA Foundation will implement the Solutions for Atrial Fibrillation Edvocacy (SAFE) demonstration project integrating atrial fibrillation (Afib) screening, detection, and referral services as a routine component of care in community-based pharmacies. The SAFE solution is designed to improve awareness about Afib, increase access to screening and education opportunities related to Afib, and offer a team-based approach to care that will ultimately improve public health outcomes.

This multi-site study will utilize community pharmacies to identify patients at-risk for Afib through point-of-care patient encounters, proactive patient profile reviews, risk assessment tools, and AliveCor's FDA-cleared EKG technology.

As part of their usual and customary care, pharmacists can identify patients potentially at-risk for Afib through routine patient encounters, proactive patient profile reviews, and subsequent discussions with the patient. Identified patients will then be asked to complete a stroke risk assessment which will help determine the patient's risk level. The pharmacist will utilize the results from the stroke risk assessment to educate the patient on why these factors could add risk, why it's important to monitor these factors, and how the patient can work to reduce or improve upon certain modifiable risk factors. All patients will be educated about the risks of Afib and the importance of future monitoring based on their risk level.

Patients will then be offered the opportunity to utilize the AliveCor EKG technology to capture an EKG reading at the point-of-care. This FDA-cleared device is easy for patients to use and a pharmacy team member will be available to guide the patient to ensure proper use. Patients who are identified as having an abnormal heart rhythm, based on their EKG reading, will be referred to their physician for evaluation and follow-up. Pharmacists will follow-up with the patients that were referred to the physician to facilitate the transition of care and inquire about confirmation of Afib and initiation of treatment. Coordination and communication among patients, pharmacists, and physicians is the foundation of this patient-centered team-based care approach.

ELIGIBILITY:
Inclusion Criteria:

* Any person at least 18 years of age
* Person who is able to present to a pharmacist for usual and customary care

Exclusion Criteria:

* Persons who are pregnant
* Persons who are lacking in capacity
* Persons who have a pacemaker or implantable cardioverter defibrillator (ICD) or other implanted electronic devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are at least 18 years of age who does not have a pacemaker or implantable cardioverter defibrillator (ICD) or other implanted electronic devices, is not pregnant, is not lacking capacity, and presenting to a pharmacist for usual and customary care.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Completion of atrial fibrillation screenings by pharmacists | September through December 2021
  Number of Afib screening tests performed in the pharmacy
Abnormal rhythm detections identified by pharmacists | September through December 2021
  Number of abnormal rhythm detections identified by AliveCor KardiaMobile technology
Physician referrals made by pharmacists | September through December 2021
  Number of physician follow-up referrals made by the pharmacist

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Bluml, Pharmacy, Principal Investigator — American Pharmacists Association Foundation
Locations (1):
- Central Study Sponsor Facility, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No